CLINICAL TRIAL: NCT03356431
Title: Comparison Between Supervised Group Exercise and Home Exercise Program for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Michele Forgiarini Saccol, Professor of Physical Therapy and Rehabilitation's Department, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 997051404
Record Dates: First submitted 2017-10-10; First posted 2017-11-29 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Exercise therapy; Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised group exercise (Experimental): The supervised exercise group will receive a lower extremity exercise treatment, under physiotherapist supervision for 60 min, two times a week (12 sessions).
  Interventions: Other: Supervised group exercise
- Home-based exercise (Experimental): For the home-based exercise group, exercises will be demonstrated to the patient with the supervision and guidance of a physiotherapist in an exercise session. These patients will perform the same exercise protocol at home at least twice a week.
  In addition to the initial session, subjects will perform further two supervised sessions (at one week and four weeks after the initial session).
  The exercise program are the same as the supervised group exercise.
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Supervised group exercise — * Quadriceps muscle isometric contraction in sitting position 1 set of 3-3 reps × 1 min hold.
  * Isotonic quadriceps contraction with resistance band 3 sets of 10 reps x 1min hold.
  * Isotonic hamstring contraction with resistance band 3 sets of 10 reps x 1min hold.
  * Sit to stand exercise during 1 min.
  * Dynamic stepping exercise (walking up and down one step/stair during 1 min).
  * Standing calf stretch 3 x 20 sec.
  * Standing quadriceps stretching 3 x 20 sec.
  * Supine hamstring stretching 3 x 20 sec.
  Other Names: Exercise therapy
  Arms: Supervised group exercise
Other: Home-based exercise — * Quadriceps muscle isometric contraction in sitting position 1 set of 3-3 reps × 1 min hold.
  * Isotonic quadriceps contraction with resistance band 3 sets of 10 reps x 1min hold.
  * Isotonic hamstring contraction with resistance band 3 sets of 10 reps x 1min hold.
  * Sit to stand exercise during 1 min.
  * Dynamic stepping exercise (walking up and down one step/stair during 1 min).
  * Standing calf stretch 3 x 20 sec.
  * Standing quadriceps stretching 3 x 20 sec.
  * Supine hamstring stretching 3 x 20 sec.
  Other Names: Exercise therapy
  Arms: Home-based exercise

SUMMARY:
Physical exercise is a widely recommended treatment modality for osteoarthritis, which can be performed through a supervised group exercise or a home exercise program. However, up to now only little research has been conducted on the home exercise program in Brazil. The objective of this study is to compare the efficacy between supervised group exercise and home exercise program in people with knee osteoarthritis. Methods: The study population consists of 46 men and woman with knee osteoarthritis aged between 40 and 65. The patients should be clinically diagnosed with knee osteoarthritis and classified in Kelgreen-Laurence grades I, II and III. Primary outcomes are the Westerm Ontário and McMaster Universities (WOMAC), Lower Extremity Functional Scale (LEFS), Pain Catastrophizing Scale (PCS), Tampa Scale for Kinesiophobia, 40-meter walk test, isometric strength of hip (abduction and adduction) and knee (flexion and extension) and postural control. The patients are randomized into 2 groups, with one group receiving 12 sessions of supervised group exercise and the other group following an exercise program at home. The program lasts 6 weeks with both groups receiving the same exercise protocol consisting of stretching, isometric and isotonic exercises for major muscle groups in both lower extremities. The Mann-Whitney U test is used to examine the Anthropometric variables. The ANOVA is used to compare outcomes before and after treatment. A value of p< 0.05 is considered to be statistically signifcant.

ELIGIBILITY:
Inclusion Criteria:

* age between 45 and 65 years;
* Kellgren-Lawrence Grade I, II and III with knee osteoarthritis determined clinically and radiographically.

Exclusion Criteria:

* history of surgery in the lower limb;
* patients who performed physiotherapy in the last six months;
* disease or disability which contraindicate the performance of the exercise training (vestibular problems, cardiorespiratory, rheumatic and neurological diseases).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Westerm Ontário and McMaster Universities | 15 min
  The Westerm Ontário and McMaster Universities (WOMAC) questionnaire is a multidimensional measure of pain, stiffness, and physical functional disability in patients with osteoarthritis. In this study we will use the Visual Analogue Scale format with 24 items and five response levels for each item (none- 0 points, mild-25, moderate-50, severe-75 or extreme-100 points). The range of the scores is function (0-1700), pain (0-500) and stiffness (0-200) and the final score of each item is obtained by dividing the final result by the number of questions of each item. The total score is obtained by adding all the items and dividing by 24. Scores range from 0 to 100 for the total WOMAC, where 0 represents the best health status and 100 the worst possible status. The higher the score, the poorer the function.

SECONDARY OUTCOMES:
Lower Extremity Functional Scale | 10 min
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. It is intended for use on adults with lower extremity conditions. The questionnaire containing five levels for each item, representing different degrees of difficulty to perform the listed activities (1- Extreme Difficulty or Unable to Perform Activity, 2- Quite a Bit of Difficulty, 3- Moderate Difficulty, 4- A Little Bit of Difficulty, 5- No Difficulty). The columns on the scale are summed to get a total score and the scores range between 0 to 80. The higher score means less functional impairment.
Pain Catastrophizing Scale (PCS) | 10 min
  This is a 13-item scale for use in assessing catastrophizing in clinical and nonclinical populations. Each PCS item is rated on a 5-point scale: 0 (not at all) to 4 (all the time). People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain. The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52. The PCS subscales are computed by summing the responses to the following items: Rumination: Sum of items 8, 9, 10, 11 Magnification: Sum of items 6, 7, 13 Helplessness: Sum of items 1, 2, 3, 4, 5, 12. Higher values representing greater catastrophizing.
Tampa Scale for Kinesiophobia | 10 min
  The Tampa Scale for Kinesiophobia (TSK) is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. Items are scored on a 4-point Likert scale with scoring possibilities ranging from 'strongly disagree' (score=1) to 'strongly agree' (score=4). This is a self-completed questionnaire and the range of scores are from 17 to 68. A total score is calculated after inversion of the individual scores of items 4, 8, 12 and 16 and then summing responses to all 17 items. Higher scores indicate an increasing degree of kinesiophobia.
40-meter walk test | 2 min
  The 40-meter walk test assesses the time it takes to walk short distances. Participants are asked to walk as quickly but as safely as possible to a mark 10 m away, return, and repeat for a total distance of 40 m. Subjects are timed for this test and data are expressed as speed. The time it takes to cover a specified distance is recorded in seconds and id measured with a stopwatch. This time is converted to a walking speed by dividing the distance covered by the time taken and is expressed as meters/second. Higher values represent better performance.
Isometric strength of hip and knee | 35 min.
  Maximal voluntary isometric contraction is measure with a hand-held dynamometer (Microfet 2m Hoogan Health Industries, West Jordan, UT, USA). Knee extension and flexion strength will be tested isometrically at 90° of knee flexion and hip abduction and aduction strength will be in tested in side-lying. Participants are instructed to perform 3 maximal voluntary isometric contractions for 5 seconds on each leg, with 10 seconds of rest between trials. The average muscle force of three repetitions will be calculated for each muscle group. The values are measured in kilogram-force and normalized to body weight (in kilograms).
Postural control | 30 min.
  Postural control is evaluated using two force platform (AMTI, model OR6-6-2000) and patients are asked to stand barefoot with one foot on each platform, arms along the sides, remaining as stable as possible looking to a point located 3 meters in front.
  All participants will be tested under four different postural conditions (eyes open, eyes closed and firm support, foam support) during three 30-s trials with one minute of rest provided between trials . The center of pressure (COP) velocity (m/s) and amplitude for medial/lateral (m/cm2) and anterior/posterior (m/cm2) directions will be analised.
Body Mass Index | 5 min.
  Body mass index (BMI) is a measure of body fat based on height and weight. BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No